CLINICAL TRIAL: NCT01229241
Title: Prospective Randomized Double-blinded Study of Systemic Pharmacokinetics of Levobupivacaine and Ropivacaine During Continuous Epidural Infusion
Brief Title: Assessment of Systemic Pharmacokinetics of Levobupivacaine and Ropivacaine During Continuous Epidural Infusion
Acronym: LEVOROPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-019393-32
Record Dates: First submitted 2010-08-16; First posted 2010-10-27 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Anesthesia; Surgery
Keywords: local anesthetic; epidural; pharmacokinetics; plasmatic concentration; epidural continuous infusion
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levobupivacaine (Other)
  Interventions: Drug: local anesthetic
- ropivacaine (Other)
  Interventions: Drug: local anesthetic

INTERVENTIONS:
Drug: local anesthetic — postoperative 48h epidural continuous infusion,
  1. ropivacaine 0,2% (250ml)+ sufentanil 0,75mcg/ml
  2. levobupivacaine 0,125% (250ml)+ sufentanil 0,75mcg/ml
  Other Names: Chriocaina; Naropina

SUMMARY:
The aim of the study is the assessment of the systemic absorption of local anesthetics during continuous epidural infusion for postoperative pain control.

DETAILED DESCRIPTION:
In literature the systemic toxicity of bupivacaine is widely demonstrated, like the minor toxicity of levobupivacaine and ropivacaine at the same anesthetic potency. The are actually no studies in humans confronting levobupivacaine and ropivacaine under the aspect of efficacy and toxicity.The aim of the study is the assessment of the systemic absorption of local anesthetics during continuous epidural infusion for postoperative pain control.

Primary outcome:

Assessment of the plasmatic equimolar concentrations of levobupivacaine and ropivacaine during continuous epidural infusion

Secondary outcome:

Assessment of the safety level of the local anesthetic (major difference between haematic concentration of the local anesthetic and neuro-cardiotoxic dose).

Difference of the analgesic efficacy between levobupivacaine and ropivacaine. Differences in collateral effects due to the local anesthetic: hypotension and sensitive block.

Prospective randomized double-blinded clinical trial

ELIGIBILITY:
Inclusion Criteria:

* ASA I or ASA II
* Scheduled for major surgery
* written informed consent

Exclusion Criteria:

* ASA III, IV
* Emergency surgery
* Recovery in intensive care unit after surgery
* habitual opioid consumption
* cognitive or mental alterations
* coagulopathy
* piastrinemia < 100.000/mm3

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of the local anesthetics in study | during 60h after surgery
  Assessment of the equivalence of the systemic exposition of levobupivacaine and ropivacaine during 48h continuous epidural infusion with in a range of 15%.Blood samples (8) will be taken for farmacological assessment of local anesthetic plasma concentrations at time (hours) 0,+3h,+6h,+12h,+24h,+48h,+54h,+60h

SECONDARY OUTCOMES:
Assessment of the pharmacological profile of the local anesthetics in study | during 60h after surgery
  Assessment of the therapeutic index (plasma concentration of the local anesthetics in study compared to those described in literature to be related to toxic effects).
Difference between the to groups (at least 25%) in terms of pain control (1 episode of VAS>4) | Pain control (VAS, VASm, rescue dose) during the 72 h postsurgery
Difference at least 20% in presentation of collateral effects between the two groups | Continuous assessment during the 72 h post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Allegri, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Unità Operativa di Anestesia e Rianimazione - Azienda Ospedaliera San Gerardo, Monza

REFERENCES:
- [Derived] Perotti L, Cusato M, Ingelmo P, Niebel TL, Somaini M, Riva F, Tinelli C, De Andres J, Fanelli G, Braschi A, Regazzi M, Allegri M. A Comparison of Differences Between the Systemic Pharmacokinetics of Levobupivacaine and Ropivacaine During Continuous Epidural Infusion: A Prospective, Randomized, Multicenter, Double-Blind Controlled Trial. Anesth Analg. 2015 Aug;121(2):348-56. doi: 10.1213/ANE.0000000000000775. PMID 25977992